CLINICAL TRIAL: NCT06677801
Title: Changes of Immune Cell Subsets During the Treatment of Lupus with Telitacicept
Brief Title: Immune Cell Subsets in SLE Patients Treated with Telitacicept
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-1010
Record Dates: First submitted 2024-10-11; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — telitacicept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant Group (Active Comparator): SLE patients treated with Telitacicept
  Interventions: Biological: Telitacicept 160mg

INTERVENTIONS:
Biological: Telitacicept 160mg — Telitacicept 160mg weekly for 24 weeks, and peripheral subtypes of immune cells will be measured at week 0, 4, 12, and 24.

SUMMARY:
This study is a single-center cohort study. Patients with SLE who met the inclusion criteria were treated with tetanercept 160 mg once a week for a total of 24 weeks, and the clinical and laboratory indicators were collected before treatment, at the 4th week, at the 12th week, and at the 24th week, and blood samples were collected for the detection of immune cell subsets.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed active SLE, who meet at least 4 of the 11 criteria for SLE revised by the United States College of Rheumatology in 1997 at the time of diagnosis;
2. Age 18~65 years old, male or female, gender ratio is not limited;
3. SLEDAI -2k score ≥ 8 points during the screening period;
4. ANA positivity as defined by a clear reference range within half a year;
5. Maintain a stable standard treatment regimen for at least 28 days prior to the date of the first dose of trial drug. Standard regimen refers to stable use of any of the following (alone or in combination): corticosteroids, antimalarials, nonsteroidal anti-inflammatory drugs (NSAIDs), other immunosuppressants or immunomodulators including azathioprine, mycophenolate (including mycophenolate mofetil, mycophenolate mofetil), cyclophosphamide, methotrexate, leflunomide, tacrolimus, and cyclosporine.
6. Understand the purpose and trial steps of this trial, and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Renal disease: severe lupus nephritis (defined as urine protein >6g/24 hours or serum creatinine >2.5mg/dL or 221μmol/L) within 8 weeks prior to randomization, or requiring active nephritis with protocol-prohibited medications, or requiring hemodialysis or receiving prednisone ≥100mg/d or equivalent corticosteroid therapy for ≥ 14 days;
2. Neurological diseases: those with central nervous system diseases caused by SLE or non-SLE within 8 weeks prior to randomization, including but not limited to epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident, encephalitis, central nervous system vasculitis, etc.;
3. Those with obvious abnormalities in laboratory examinations: a. ALT or AST≥2×ULN (upper limit of normal); b. Endogenous creatinine clearance < 30 mL/min; c. White blood cell count < 2.5×10 9/L; d. Hemoglobin <85g/L; Platelet count < 50×10 9/L;
4. Current active hepatitis or previous severe liver lesions or medical history. Hepatitis B: excludes patients who are HBsAg positive. Patients who are HBsAg negative but HBcAb positive will need to be accounted for by HBV-DNA testing: if HBV-DNA is positive, the patient is excluded from participating in the study; If HBV-DNA is negative, the patient can participate in the study. Hepatitis C: excludes patients who are positive for hepatitis C antibodies;
5. Immunodeficiency or active infection (such as herpes zoster, HIV virus infection, active tuberculosis, etc.) during the screening period;
6. Patients with other connective tissue diseases, history of malignancy, or active/recurrent peptic ulcer;
7. Pregnant women, lactating women, and males or females with birth plans during the trial;
8. Those who have received a live vaccine within 28 days prior to randomization;
9. Participation in any clinical trial within 28 days prior to randomization or within 5 times the half-life of the investigational drug enrolled in the clinical trial (whichever is longer);
10. Use of B-cell-targeted therapy agents such as rituximab, epacizumab or belimumab, etc., within 12 months prior to randomization;
11. Use of tumor necrosis factor inhibitors, interleukin receptor blockers within 12 months prior to randomization;
12. Those who have been treated with intravenous immunoglobulin (IVIG), prednisone ≥ 100mg/d, or equivalent corticosteroids for ≥ 14 days within 28 days prior to randomization, and those who have undergone plasmapheresis;
13. Use of interleukin-2, thalidomide, tripterygium wilfordii and tripterygium wilfordii-containing traditional Chinese medicine preparations within 28 days prior to randomization;
14. Allergic reactions: history of allergy to human-derived biological products;
15. Mentally ill persons with depression or suicidal thoughts;
16. Those who are considered inappropriate by the investigator to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes of immune cell subsets after treatment | 24 weeks

SECONDARY OUTCOMES:
SLE responder index (SRI) -4 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China